CLINICAL TRIAL: NCT03949569
Title: A Pilot Study of the Effects of Interactions With Therapy Dogs on Child Stress Responsivity
Brief Title: The Effects of Therapy Dogs on Child Biology and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB18-0472; R21HD094956 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-05-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Stress Reaction; Behavior, Social
Keywords: Children; Human-Animal Interaction; Stress; Cortisol
MeSH Terms: conditions — Fractures, Stress; Social Behavior; Human-Animal Interaction

STUDY DESIGN:
Intervention Model Description: The investigators will use a randomized crossover design. All children will receive two interventions during a single study visit. Children will be assigned to one of three research design arms using a stratified random sampling approach with child sex balanced across arm (N=110 in each group). All children will participate in the same tasks, in the same order. The only difference between research design arms is the timing of the interventions. In one arm the child will interact with the therapy dog prior to the psychosocial stress test and will interact with the stuffed toy dog prior to the behavioral tasks; the reverse is true for children in the second arm. In the third arm, the child will watch a 5 minute puppy video prior to the psychosocial stress test and will interact with the stuffed toy dog prior to the behavioral tasks
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be unaware of which study arm they are assigned. Individuals performing the interventions will be blind to study condition. The investigator will be blind to study condition until data analysis. Video data will be coded by observers blind to the study condition. The primary outcomes assessor is not blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): In this condition, children will interact with the therapy dog prior to the psychosocial stress task and with the stuffed toy dog prior to the prosocial behavior tests.
  Interventions: Behavioral: Therapy Dog; Behavioral: Stuffed Toy Dog
- Arm 2 (Experimental): In this condition, children will interact with the stuffed toy prior to the psychosocial stress task collection and with the therapy dog prior to the prosocial behavior tests.
  Interventions: Behavioral: Therapy Dog; Behavioral: Stuffed Toy Dog
- Arm 3 (Experimental): In this condition, children will watch a 5 minute puppy video prior to the psychosocial stress task collection and with the therapy dog prior to the prosocial behavior tests.
  Interventions: Behavioral: Stuffed Toy Dog; Behavioral: 5 Minute Puppy Video

INTERVENTIONS:
Behavioral: Therapy Dog — Children will undergo a 5 minute unstructured session with either a certified therapy dog or with a dog who is trained and certified for animal-assisted interventions and/or animal-assisted activities. Children will be allowed to talk to, pet, and play with the therapy dog during the interaction.
  Arms: Arm 1; Arm 2
Behavioral: Stuffed Toy Dog — Children will undergo a 5 minute unstructured session with a stuffed toy dog. Children will be allowed to talk to, pet, and play with the stuffed toy dog during the interaction.
Behavioral: 5 Minute Puppy Video — Children will watch a 5 minute puppy video.
  Arms: Arm 3

SUMMARY:
The objective of this study is to apply a rigorous experimental design to test whether children's interactions with therapy dogs increase immediate prosocial behavior and reduce immediate biological response to stress.

DETAILED DESCRIPTION:
The central goal of the study is to determine whether brief interactions with a therapy dog have an immediate impact on children's biological response to stress, prosocial behaviors, and self-reported mood in comparison to interactions with a stuffed toy dog. The study uses a randomized crossover design with two study arms; all children will receive the both interventions during the same session, with the timing of the intervention randomized across subject. All outcomes will be assessed during a single study visit. No follow-up data will be collected.

The study uses both between-group and within-subject comparisons. Between groups, the investigators predict that children who interact with a therapy dog prior to a psychosocial stress task (Arm 1) will show attenuated cortisol response to the stress task (primary outcome) and reduced physiological stress (secondary outcomes) compared to children who interact with a stuffed toy dog prior to the psychosocial stress task (Arm 2). As an additional control, children will also watch a 5 minute puppy video prior to the prosocial stress task and will then interact with a stuffed toy dog prior to the psychosocial stress task (Arm 3).

Conversely, children who interact with the therapy dog immediately prior to the in-lab behavior tasks (Arm 2) will show higher levels of behavioral carefulness and prosocial behavior (primary outcomes) compared to children who interact with the stuffed toy dog prior to the behavior tasks (Arm 1).

Within subjects across both study arms, increases in positive mood and decreases in negative mood (secondary outcomes) will be greatest following interaction with the therapy dog compared to the stuffed toy dog, after controlling for main effects of study arm. Within subjects, physiological markers of stress (secondary outcomes) will be lower during the interaction with the therapy dog than during interaction with the stuffed toy dog.

Investigators will seek additional funds to collect and analyze salivary oxytocin data. The hypothesis is that children will show greater increase in oxytocin following interaction with the therapy dog in comparison to interaction with the stuffed toy dog.

This study will also investigate the mechanisms through which child-dog interactions influence youth stress responsivity, using coded videotaped data from the subset of children in Arm 1 who interact with the therapy dog prior to the psychosocial stress task. It is hypothesized that child behaviors observed during the interaction, such as duration and frequency of eye gaze, petting and stroking behaviors, and use of positive affect, will be inversely correlated with change in cortisol response to stress. Dog behaviors, such as duration and frequency of eye gaze and approach behaviors, will be inversely correlated with children's change in cortisol response to stress.

The study will also investigate whether child characteristics moderate the effects of the child-dog interaction. Investigators hypothesize that the effects of the therapy dog intervention will be stronger among children who currently live with dogs versus non-dog owning children and among children with more positive attitudes towards pets. It is also expected that the effects of the therapy dog interaction will be weaker among children with internalizing problems and for children experiencing higher levels of general stress. Investigators will also test whether the effects of the therapy dog intervention vary across child gender, race/ethnicity, or socioeconomic status, or child personality.

ELIGIBILITY:
Inclusion Criteria:

- Children between the ages of 8-12 years old

Exclusion Criteria:

* Limited comprehension of English
* Severe neurological, medical, or psychiatric illnesses (e.g., schizophrenia, psychosis)
* Severe asthma or animal allergies
* Animal phobias
* Use of medications that affect cortisol

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Mean level and Change in Salivary cortisol | Measured at baseline and over a 45 minute period before and after the psychosocial stress test
  Salivary cortisol will be collected 7 times during the study visit.
Mean level Prosocial behavior assessed with the Zurich prosocial game | Assessed after the 2nd intervention.
  During the study visit prosocial behavior is assessed through total number of helping behaviors recorded during the Zurich prosocial game.
Mean level Behavioral carefulness assessed with the children's game, Operation | Assessed after the 2nd intervention.
  During the study visit, participants will play the game Operation. Behavioral carefulness metrics include number of errors and total time to complete the task.

SECONDARY OUTCOMES:
Mean level and Change in Psychological Well Being assessed by the Positive and Negative Affect Scale for Children (PANAS-C) | Measured at the beginning of the study visit and before and after each intervention.
  The PANAS-C will be administered repeatedly during the study visit.
Mean level and Change in galvanic skin response measured with the E4 wristband | Assessed during both interventions and during the psychosocial stress test.
  Participants will wear an E4 wristband during the study visit that records continuous physiological markers of stress.
Mean level and Change in heart rate measured with the E4 wristband | Assessed during both interventions and during the psychosocial stress test.
  Participants will wear an E4 wristband during the study visit that records continuous physiological markers of stress.

OTHER OUTCOMES:
Mean Level and Change in Salivary Oxytocin (pending additional funds) | Assessed immediately before and after each intervention.
  Salivary oxytocin will be measured repeatedly during the study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen C Jacobson, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying research publications
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after publication and will be available for up to 5 years post-publication.
Access Criteria: The PI will evaluate written requests for IPD sharing. All requests must be made from individuals with legitimate research questions and must be compliant with IRB regulations.

REFERENCES:
- [Background] Merikangas KR, He JP, Brody D, Fisher PW, Bourdon K, Koretz DS. Prevalence and treatment of mental disorders among US children in the 2001-2004 NHANES. Pediatrics. 2010 Jan;125(1):75-81. doi: 10.1542/peds.2008-2598. Epub 2009 Dec 14. PMID 20008426
- [Background] Costello EJ, Egger H, Angold A. 10-year research update review: the epidemiology of child and adolescent psychiatric disorders: I. Methods and public health burden. J Am Acad Child Adolesc Psychiatry. 2005 Oct;44(10):972-86. doi: 10.1097/01.chi.0000172552.41596.6f. PMID 16175102
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Lewinsohn PM, Zinbarg R, Seeley JR, Lewinsohn M, Sack WH. Lifetime comorbidity among anxiety disorders and between anxiety disorders and other mental disorders in adolescents. J Anxiety Disord. 1997 Jul-Aug;11(4):377-94. doi: 10.1016/s0887-6185(97)00017-0. PMID 9276783
- [Background] Kessler RC, Petukhova M, Sampson NA, Zaslavsky AM, Wittchen H -U. Twelve-month and lifetime prevalence and lifetime morbid risk of anxiety and mood disorders in the United States. Int J Methods Psychiatr Res. 2012 Sep;21(3):169-84. doi: 10.1002/mpr.1359. Epub 2012 Aug 1. PMID 22865617
- [Background] Kiecolt-Glaser JK, McGuire L, Robles TF, Glaser R. Emotions, morbidity, and mortality: new perspectives from psychoneuroimmunology. Annu Rev Psychol. 2002;53:83-107. doi: 10.1146/annurev.psych.53.100901.135217. PMID 11752480
- [Background] Miller GE, Chen E, Parker KJ. Psychological stress in childhood and susceptibility to the chronic diseases of aging: moving toward a model of behavioral and biological mechanisms. Psychol Bull. 2011 Nov;137(6):959-97. doi: 10.1037/a0024768. PMID 21787044
- [Background] Adam EK, Kumari M. Assessing salivary cortisol in large-scale, epidemiological research. Psychoneuroendocrinology. 2009 Nov;34(10):1423-36. doi: 10.1016/j.psyneuen.2009.06.011. Epub 2009 Jul 31. PMID 19647372
- [Background] Sapolsky RM, Romero LM, Munck AU. How do glucocorticoids influence stress responses? Integrating permissive, suppressive, stimulatory, and preparative actions. Endocr Rev. 2000 Feb;21(1):55-89. doi: 10.1210/edrv.21.1.0389. PMID 10696570
- [Background] McEwen BS. Stress, adaptation, and disease. Allostasis and allostatic load. Ann N Y Acad Sci. 1998 May 1;840:33-44. doi: 10.1111/j.1749-6632.1998.tb09546.x. PMID 9629234
- [Background] Gunnar MR, Quevedo KM. Early care experiences and HPA axis regulation in children: a mechanism for later trauma vulnerability. Prog Brain Res. 2008;167:137-49. doi: 10.1016/S0079-6123(07)67010-1. PMID 18037012
- [Background] Miller GE, Chen E, Zhou ES. If it goes up, must it come down? Chronic stress and the hypothalamic-pituitary-adrenocortical axis in humans. Psychol Bull. 2007 Jan;133(1):25-45. doi: 10.1037/0033-2909.133.1.25. PMID 17201569
- [Background] Klein ZA, Romeo RD. Changes in hypothalamic-pituitary-adrenal stress responsiveness before and after puberty in rats. Horm Behav. 2013 Jul;64(2):357-63. doi: 10.1016/j.yhbeh.2013.01.012. Epub 2013 Mar 7. PMID 23465865
- [Background] Lightman SL. The neuroendocrinology of stress: a never ending story. J Neuroendocrinol. 2008 Jun;20(6):880-4. doi: 10.1111/j.1365-2826.2008.01711.x. PMID 18601712
- [Background] Costello EJ, He JP, Sampson NA, Kessler RC, Merikangas KR. Services for adolescents with psychiatric disorders: 12-month data from the National Comorbidity Survey-Adolescent. Psychiatr Serv. 2014 Mar 1;65(3):359-66. doi: 10.1176/appi.ps.201100518. PMID 24233052
- [Background] Sobo EJ, Eng B, Kassity-Krich N. Canine visitation (pet) therapy: pilot data on decreases in child pain perception. J Holist Nurs. 2006 Mar;24(1):51-7. doi: 10.1177/0898010105280112. PMID 16449747
- [Background] Braun C, Stangler T, Narveson J, Pettingell S. Animal-assisted therapy as a pain relief intervention for children. Complement Ther Clin Pract. 2009 May;15(2):105-9. doi: 10.1016/j.ctcp.2009.02.008. Epub 2009 Mar 3. PMID 19341990
- [Background] Crossman MK. Effects of Interactions With Animals On Human Psychological Distress. J Clin Psychol. 2017 Jul;73(7):761-784. doi: 10.1002/jclp.22410. Epub 2016 Nov 3. PMID 27809353
- [Background] Cohen SP. Can pets function as family members? West J Nurs Res. 2002 Oct;24(6):621-38. doi: 10.1177/019394502320555386. PMID 12365764
- [Background] Allen KM, Blascovich J, Tomaka J, Kelsey RM. Presence of human friends and pet dogs as moderators of autonomic responses to stress in women. J Pers Soc Psychol. 1991 Oct;61(4):582-9. doi: 10.1037//0022-3514.61.4.582. PMID 1960650
- [Background] Polheber JP, Matchock RL. The presence of a dog attenuates cortisol and heart rate in the Trier Social Stress Test compared to human friends. J Behav Med. 2014 Oct;37(5):860-7. doi: 10.1007/s10865-013-9546-1. Epub 2013 Oct 30. PMID 24170391
- [Background] Allen K, Blascovich J, Mendes WB. Cardiovascular reactivity and the presence of pets, friends, and spouses: the truth about cats and dogs. Psychosom Med. 2002 Sep-Oct;64(5):727-39. doi: 10.1097/01.psy.0000024236.11538.41. PMID 12271103
- [Background] Kertes DA, Liu J, Hall NJ, Hadad NA, Wynne CDL, Bhatt SS. Effect of Pet Dogs on Children's Perceived Stress and Cortisol Stress Response. Soc Dev. 2017 May;26(2):382-401. doi: 10.1111/sode.12203. Epub 2016 Jul 28. PMID 28439150
- [Background] Odendaal JS, Meintjes RA. Neurophysiological correlates of affiliative behaviour between humans and dogs. Vet J. 2003 May;165(3):296-301. doi: 10.1016/s1090-0233(02)00237-x. PMID 12672376
- [Background] Barker SB, Knisely JS, McCain NL, Best AM. Measuring stress and immune response in healthcare professionals following interaction with a therapy dog: a pilot study. Psychol Rep. 2005 Jun;96(3 Pt 1):713-29. doi: 10.2466/pr0.96.3.713-729. PMID 16050629
- [Background] Viau R, Arsenault-Lapierre G, Fecteau S, Champagne N, Walker CD, Lupien S. Effect of service dogs on salivary cortisol secretion in autistic children. Psychoneuroendocrinology. 2010 Sep;35(8):1187-93. doi: 10.1016/j.psyneuen.2010.02.004. Epub 2010 Mar 1. PMID 20189722
- [Background] Beetz A, Julius H, Turner D, Kotrschal K. Effects of social support by a dog on stress modulation in male children with insecure attachment. Front Psychol. 2012 Sep 28;3:352. doi: 10.3389/fpsyg.2012.00352. eCollection 2012. PMID 23162482
- [Background] Redefer LA, Goodman JF. Brief report: pet-facilitated therapy with autistic children. J Autism Dev Disord. 1989 Sep;19(3):461-7. doi: 10.1007/BF02212943. No abstract available. PMID 2793790
- [Background] Martin F, Farnum J. Animal-assisted therapy for children with pervasive developmental disorders. West J Nurs Res. 2002 Oct;24(6):657-70. doi: 10.1177/019394502320555403. PMID 12365766
- [Background] Nagasawa M, Kikusui T, Onaka T, Ohta M. Dog's gaze at its owner increases owner's urinary oxytocin during social interaction. Horm Behav. 2009 Mar;55(3):434-41. doi: 10.1016/j.yhbeh.2008.12.002. Epub 2008 Dec 14. PMID 19124024
- [Background] Westgarth C, Heron J, Ness AR, Bundred P, Gaskell RM, Coyne KP, German AJ, McCune S, Dawson S. Family pet ownership during childhood: findings from a UK birth cohort and implications for public health research. Int J Environ Res Public Health. 2010 Oct;7(10):3704-29. doi: 10.3390/ijerph7103704. Epub 2010 Oct 18. PMID 21139856
- [Background] Risley-Curtiss C, Holley LC, Wolf S. The animal-human bond and ethnic diversity. Soc Work. 2006 Jul;51(3):257-68. doi: 10.1093/sw/51.3.257. PMID 17076123
- [Background] Sable P. Pets, attachment, and well-being across the life cycle. Soc Work. 1995 May;40(3):334-41. PMID 7761919
- [Background] McBurnett K, Lahey BB, Frick PJ, Risch C, Loeber R, Hart EL, Christ MA, Hanson KS. Anxiety, inhibition, and conduct disorder in children: II. Relation to salivary cortisol. J Am Acad Child Adolesc Psychiatry. 1991 Mar;30(2):192-6. doi: 10.1097/00004583-199103000-00005. PMID 2016221
- [Background] Badanes LS, Watamura SE, Hankin BL. Hypocortisolism as a potential marker of allostatic load in children: associations with family risk and internalizing disorders. Dev Psychopathol. 2011 Aug;23(3):881-896. doi: 10.1017/S095457941100037X. PMID 21756439
- [Background] Davis EP, Donzella B, Krueger WK, Gunnar MR. The start of a new school year: individual differences in salivary cortisol response in relation to child temperament. Dev Psychobiol. 1999 Nov;35(3):188-96. doi: 10.1002/(sici)1098-2302(199911)35:33.0.co;2-k. PMID 10531531
- [Background] Spies LA, Margolin G, Susman EJ, Gordis EB. Adolescents' cortisol reactivity and subjective distress in response to family conflict: the moderating role of internalizing symptoms. J Adolesc Health. 2011 Oct;49(4):386-92. doi: 10.1016/j.jadohealth.2011.01.014. Epub 2011 Jun 2. PMID 21939869
- [Background] Dockray S, Susman EJ, Dorn LD. Depression, cortisol reactivity, and obesity in childhood and adolescence. J Adolesc Health. 2009 Oct;45(4):344-50. doi: 10.1016/j.jadohealth.2009.06.014. Epub 2009 Aug 3. PMID 19766938
- [Background] Virues-Ortega J, Buela-Casal G. Psychophysiological effects of human-animal interaction: theoretical issues and long-term interaction effects. J Nerv Ment Dis. 2006 Jan;194(1):52-7. doi: 10.1097/01.nmd.0000195354.03653.63. PMID 16462556
- [Background] Havener L, Gentes L, Thaler B, Megel ME, Baun MM, Driscoll FA, Beiraghi S, Agrawal S. The effects of a companion animal on distress in children undergoing dental procedures. Issues Compr Pediatr Nurs. 2001 Apr-Jun;24(2):137-52. doi: 10.1080/01460860118472. PMID 11817428
- [Background] Avenevoli S, Swendsen J, He JP, Burstein M, Merikangas KR. Major depression in the national comorbidity survey-adolescent supplement: prevalence, correlates, and treatment. J Am Acad Child Adolesc Psychiatry. 2015 Jan;54(1):37-44.e2. doi: 10.1016/j.jaac.2014.10.010. Epub 2014 Oct 29. PMID 25524788
- [Background] Cummings JR, Druss BG. Racial/ethnic differences in mental health service use among adolescents with major depression. J Am Acad Child Adolesc Psychiatry. 2011 Feb;50(2):160-70. doi: 10.1016/j.jaac.2010.11.004. Epub 2010 Dec 31. PMID 21241953
- [Background] Smalley KB, Yancey CT, Warren JC, Naufel K, Ryan R, Pugh JL. Rural mental health and psychological treatment: a review for practitioners. J Clin Psychol. 2010 May;66(5):479-89. doi: 10.1002/jclp.20688. PMID 20222125
- [Background] Leiberg S, Klimecki O, Singer T. Short-term compassion training increases prosocial behavior in a newly developed prosocial game. PLoS One. 2011 Mar 9;6(3):e17798. doi: 10.1371/journal.pone.0017798. PMID 21408020
- [Background] Gunnar MR, Talge NM, Herrera A. Stressor paradigms in developmental studies: what does and does not work to produce mean increases in salivary cortisol. Psychoneuroendocrinology. 2009 Aug;34(7):953-67. doi: 10.1016/j.psyneuen.2009.02.010. Epub 2009 Mar 24. PMID 19321267
- [Background] Eisenberg N, Fabes RA, Schaller M, Miller P, Carlo G, Poulin R, Shea C, Shell R. Personality and socialization correlates of vicarious emotional responding. J Pers Soc Psychol. 1991 Sep;61(3):459-70. PMID 1941517
- [Background] Luby JL, Svrakic DM, McCallum K, Przybeck TR, Cloninger CR. The Junior Temperament and Character Inventory: preliminary validation of a child self-report measure. Psychol Rep. 1999 Jun;84(3 Pt 2):1127-38. doi: 10.2466/pr0.1999.84.3c.1127. PMID 10477935
- [Background] Sherman GD, Haidt J, Coan JA. Viewing cute images increases behavioral carefulness. Emotion. 2009 Apr;9(2):282-6. doi: 10.1037/a0014904. PMID 19348541
- [Background] Belli RF. The structure of autobiographical memory and the event history calendar: potential improvements in the quality of retrospective reports in surveys. Memory. 1998 Jul;6(4):383-406. doi: 10.1080/741942610. PMID 9829098
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417